CLINICAL TRIAL: NCT02587169
Title: GEIS-27: Phase I/II Multicenter and Prospective Trial of Nilotinib and Adriamycin as Neoadjuvant Treatment in Liposarcomas and Leiomyosarcomas of Retroperitoneum
Brief Title: Trial of Nilotinib and Adriamycin as Treatment in Liposarcomas and Leiomyosarcomas of Retroperitoneum
Acronym: GEIS-27
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Broto, Javier Martín, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC10-150 RETRONEO; 2011-002368-26 (EudraCT Number); GEIS-27 (Other: Spanish Sarcoma Group (GEIS))
Record Dates: First submitted 2013-07-17; First posted 2015-10-27 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Retroperitoneal Liposarcoma; Retroperitoneal Leiomyosarcoma; Chondrosarcoma
Keywords: liposarcoma; leiomyosarcoma; retroperitoneum; chondrosarcoma
MeSH Terms: conditions — Retroperitoneal liposarcoma; Chondrosarcoma; Liposarcoma; Leiomyosarcoma | interventions — nilotinib; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nilotinib-adriamycin (Experimental): The nilotinib-adriamycin combination will be given in 4 cycles of 21 days. In each cycle, nilotinib will be administered at fixed dose of 400 mg/12h orally during 6 consecutive days (1-6) and endovenous adriamycin (20 minutes) on day 5 at three levels (in phase I, dosage of 60 mg/m2, 65 mg/m2, and 75 mg/m2 will be tested to determine the recommended dose for phase II).
  Interventions: Drug: Nilotinib-adriamycin

INTERVENTIONS:
Drug: Nilotinib-adriamycin — The nilotinib-adriamycin combination will be given in 4 cycles of 21 days. In each cycle, nilotinib will be administered at fixed dose of 400 mg/12h orally during 6 consecutive days (1-6) and endovenous adriamycin (20 minutes) on day 5 at three levels (in phase I, dosage of 60 mg/m2, 65 mg/m2, and 75 mg/m2 will be tested to determine the recommended dose for phase II).
  Other Names: Nilotinib Tasigna; Doxorubicin hydrochloride

SUMMARY:
Phase I/II multicenter and prospective trial of nilotinib and adriamycin as neoadjuvant treatment in liposarcomas and leiomyosarcomas of retroperitoneum.

The main objective of this study is to improve relapse-free survival (RFS)and overall survival (OS) decreasing from 50% to 30% the relapse percentage at 5 years in patients with resected sarcoma of retroperitoneum.

Secondary objectives include the analysis of antitumoral activity through response rate (RECIST and tissular changes), the assessment of positive correlation between biomarkers and clinical results, the study of long term overall survival, and the analysis of the safety profile of the nilotinib-adriamycin combination.

The trial hypothesis is that the nilotinib-adriamycin combination is synergistic and therefore better response results are expected (from 20% as P0 to 40% as P1). The study seeks to find a positive correlation between biomarkers and clinical results in retroperitoneal liposarcoma and leiomyosarcoma treated with the mentioned combination.

The study involves the participation of 20 hospitals of the Spanish Sarcoma Group (GEIS). The treatment consists of 4 neoadjuvant cycles of nilotinib-adriamycin on patients with resectable retroperitoneal sarcoma. The research comprises a robust translational study as well as histological and radiological reviews.

DETAILED DESCRIPTION:
The nilotinib-adriamycin combination will be given in 4 cycles of 21 days. In each cycle, nilotinib will be administered at fixed dose of 400 mg/12h orally during 6 consecutive days (1-6) and endovenous adriamycin (20 minutes) on day 5 at three levels (in phase I, dosage of 60 mg/m2, 65 mg/m2, and 75 mg/m2 will be tested to determine the recommended dose for phase II).

Phase I includes patients with retroperitoneal liposarcoma, retroperitoneal leiomyosarcoma and chondrosarcoma. Phase II is focused on retroperitoneal liposarcoma and leiomyosarcoma only.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological diagnosis of well differentiated liposarcoma, dedifferentiated liposarcoma or primary leiomyosarcoma of retroperitoneum and resectable. In phase I the study will recruit patients with high-grade chondrosarcoma of non-mesenchymal type.
* Age: 18-70 years.
* Measurable disease, according to RECIST criteria.
* Functional status: 0-1 (ECOG).
* Baseline medullar function (hemoglobin > 10 g/dL, leukocytes ≥ 3.000/mm3, RAN≥ 1,5 x 109 /l, granulocytes ≥ 1.500/mm3, platelets ≥ 100.000/mm3). Patients with alteration of transaminases ≤ 2.5 times the normal limits, bilirubin total ≤ LSN, CPK≤ 2.5 times the normal limits, alkaline phosphatase ≤ 2.5 times more the normal limits or creatinine values ≤ 1.6 mg/dL, are accepted.
* Cardiac function (LVEF) normal, considering the normal ranges of the institution.
* The patient must voluntarily sign the informed consent before any trial test, knowing that he/she can leave the trial at any time, without any consequence for his/her posterior medical attention.
* Patients in fertile age (both male and female) must use an effective contraceptive method before the entry in the study and during the trial. Moreover, women must maintain contraceptive measures up to 5 months after the treatment. Pregnancy must be ruled out though urine test (negative pregnancy test) for study enrolment.

Exclusion Criteria:

* Patients having received previous chemotherapy.
* Patient having been irradiated on the tumoral disease.
* Functional status > 1 (ECOG).
* Metastasis in any location.
* Bilirubin values over the normal level. Creatinine over 1.6 mg/dL.
* History of another oncological disease except basalioma or in situ cervical carcinoma adequately treated.
* Serious cardiovascular diseases (dyspnea >= 2 NYHA, ie.)
* Systemic pathologies limiting survival to less than 2 years, limiting patient availability, or those that, by clinical judgement, may interfere significantly with treatment toxicity.
* Bacterial, viral, or uncontrolled mycotic infectious diseases.
* Pregnant or lactating patients.
* Psychological, family, sociological or geographical situations not allowing protocol fulfilment or informed consent signature.
* Patients currently involved in other clinical trials receiving any other agent under investigation.
* Patient having participated in a clinical trial and/or having received an agent under investigation in the 30 days prior to enrolment.
* Patients requiring treatments with prolongation of QT interval as amiodarone, disopyramide, procainamide, quinidine, and sotalol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival (RFS) at 5 years | 5 years
  The main goal of the study is to improve relapse-free survival (RFS) and overall survival (OS) decreasing from 50% to 30% the percentage of relapse at 5 years in patients with resected retroperitoneal sarcoma.

SECONDARY OUTCOMES:
Objective response rate (ORR) (confirmed complete response [CR] and partial response [PR]) | Baseline and at 4 months
  To determine the objective response rate (ORR) (confirmed complete response [CR] and partial response [PR]) using RECIST 1.1 criteria
Overall survival (OS) | 100 months
  Overall survival measured from treatment start date until date of death, whichever the cause, assessed up to 100 months
Number of adverse events | 4 months
  Number and type of adverse events according to CTCAE 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Javier Martín, MD, PhD, Study Director — Spanish Sarcoma Group (GEIS)
Locations (20):
- Spain (20):
  - Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Infanta Cristina, Badajoz
  - Hospital Universitari Germans Trials i Pujol, Badalona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Provincial de Castellón, Castellon
  - Complejo Asistencial Universitario de León, León
  - Hospital Puerta de Hierro, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Marqués de Valdecilla, Santander
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela
  - Hospital Virgen del Rocío, Seville
  - Hospital Virgen de la Salud, Toledo
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Xeral Cies, Vigo
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- See also: Spanish Sarcoma Group (GEIS) — http://www.grupogeis.org